CLINICAL TRIAL: NCT01063218
Title: Phase IV - Evaluation of Cetaphil Advanced Usage to Control Light to Moderate Atopic Dermatitis, in Attempt to Reduce the Necessity of Topic Corticoids Application
Brief Title: Evaluation of Cetaphil Advanced Usage to Control Light to Moderate Atopic Dermatitis, in Attempt to Reduce the Necessity of Topic Corticoids Application
Status: Completed | Phase: Phase 4 | Type: Interventional
Sponsor: Galderma Brasil Ltda. (Industry)
Responsible Party: Mario Cézar Pires, Complexo Hospitalar Padre Bento de Guarulhos
Allocation: Non-Randomized | Model: Single Group | Masking: None | Purpose: Prevention
Other Study IDs: BR.09.001
Record Dates: First submitted 2010-02-04; First posted 2010-02-05 (Estimated); Last update posted 2012-03-12 (Estimated); Status verified 2012-03

CONDITIONS: Dermatitis, Atopic
Keywords: Dermatitis, Atopic; Corticoids, topic; Corticosteroids
MeSH Terms: conditions — Dermatitis, Atopic

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (1):
- Emollient (Other): Only one arm: Emollient (Cetaphil Advanced) to be applied twice a day
  Interventions: Other: Emollient - Cetaphil Advanced

INTERVENTIONS:
Other: Emollient - Cetaphil Advanced — Emollient - Cetaphil Advanced - to be applied twice a day for 20 weeks.

SUMMARY:
The main goal of this present study is evaluate the decreasing of necessity of topic corticoids usage to control outbreaks of light to moderate atopic dermatitis by using the correct emollients.

ELIGIBILITY:
Inclusion Criteria:

* Male or Female patients
* 2 to 10 years old.
* with light to moderate with no signs of acute/ sub-acute eczema or in activity.
* Subjects can not present inflammatory lesions, erythema, edema, eschar, excoriation and lichens.
* Subjects can present light to moderate dryness.

Exclusion Criteria:

* Subjects presenting any serious systemic disease
* Subjects with medical history regarding serious asthma
* Subjects with known or suspected allergy to one of the investigational products
* Subjects with acute atopic eczema or in activity, needing systemic antibiotics
* Subjects with signs of active infections on skin
* Subjects whose parents or legal guardian seem to have difficulty in understand the informed consent form (ICF)
* Female subjects who are not in pre-menarche period.
* Subjects who need topic corticoids or any other medication that can interfere on Atopic Dermatitis during the study.
* Patient with a wash-out period for treatment less than:
* injectable corticoids: 60 days
* systemic corticoids: 15 days
* topic corticoids: 8 days
* topic immunomodulator: 8 days
* antihistaminic : 48 hours

Ages: 2 Years to 10 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Child
Enrollment: 74 (Estimated)
Dates: Start 2009-12; Primary Completion 2010-09 (Actual); Study Completion 2010-10 (Actual)

PRIMARY OUTCOMES:
clinical evaluation | Baseline, Weeks 2, 4, 6, 8, 10, 12, 16, 20 and 24

CONTACTS AND LOCATIONS:
Overall Officials: Mario C Pires, MD, Principal Investigator — Complexo Hospitalar Padre Bento de Guarulhos; Izelda Costa, MD, Principal Investigator — Hospital Universitário de Brasília
Locations (2):
- Brazil (2):
  - Hospital Universitário de Brasília, Brasília, Federal District
  - Complexo Hospitalar Padre Bento de Guarulhos, Guarulhos, São Paulo